CLINICAL TRIAL: NCT03427567
Title: A Multi-centre Real-world Non-interventional Observational Study to Evaluate Effectiveness of Sublobar Dissection in the Chinese Patients With Non-small Cell Lung Cancer
Brief Title: A Study to Evaluate Effectiveness of Sublobar Dissection in Patients With Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, XiangNing Fu, Professor, Tongji Hospital
Other Study IDs: TJ-LC-01
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Chinese; real-world evidences; NSCLC; sublobar dissection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sublobar dissection: Chinese NSCLC patients who received sublobar dissection
  Interventions: Procedure: Sublobar dissection

INTERVENTIONS:
Procedure: Sublobar dissection — Sublobar dissection plus lymphadenectomy
  Other Names: Surgeries

SUMMARY:
A study to evaluate effectiveness of sublobar dissection in patients with non-small cell lung cancer

DETAILED DESCRIPTION:
This is a multi-centre real-world non-interventional observational study. The study data on patient demographic/tumor biological characteristics and clinical treatments were retrospectively collected to evaluate effectiveness of sublobar dissection in the Chinese patients with non-small cell lung cancer who received sublobar dissection.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old;
* Patients who received sublobar dissection from 2014 to 2017 (segment dissection/wedge dissection/segment and wedge dissections);
* Patients who received selective or systematic lymphadenectomy;
* Pathologically diagnosed patients with non-small cell lung cancer;
* Pathological staging: I, II

Exclusion Criteria:

* Patients who received cancer treatments before surgeries (adjuvant therapies including chemotherapies, radiotherapies, target therapies);
* Patients who received late-phase or intolerant palliative lobectomy or compromise sublobar dissection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with pathological diagnosed non-small cell lung cancer who received sublobar dissection and lymphadenectomy
Sampling Method: Non-Probability Sample
Enrollment: 3902 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2014 - 2017
  Overall survival

SECONDARY OUTCOMES:
Overall survivals in subgroups | 2014 - 2017
  Overall survivals categorised by tumor biological characteristics

OTHER OUTCOMES:
Impact factors of overall survival | 2014 - 2017
  Impact factors of overall survival as measured by patient demographic/tumor biological characteristics and clinical treatments
Death rates after surgeries | 2014 - 2017
  Death rates after surgeries
Impact factors of death rates after surgeries | 2014 - 2017
  Impact factors of death rates after surgeries
Incidence of complications after surgeries | 2014 - 2017
  Incidence of complications after surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Xiangning Fu, PhD, Principal Investigator — Tongji Hospital Affiliated to Tongji Medical College Huazhong Technology University
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan cancer hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No